CLINICAL TRIAL: NCT06087770
Title: An Open-label, Dose-escalation Phase Ia Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of SM3321 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Clinical Study of SM3321 With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing StarMab Biomed Technology Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SM3321-CN-001
Record Dates: First submitted 2023-08-03; First posted 2023-10-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: locally advanced; solid tumors; metastatic
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase Ia Dose escalation (Experimental): Phase Ia Dose escalation： A maximum of 48 patients will be enrolled in this phase and are planned to be divided into eight dose groups: 0.3 mg/kg, 1mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg, 40 mg/kg and 50 mg/kg
  Interventions: Drug: SM3321

INTERVENTIONS:
Drug: SM3321 — Intravenous infusion, once a week, 28 days for a dosing cycle

SUMMARY:
The purpose of this study is to evaluate the Safety and Tolerability of SM3321 in patients with locally advanced or metastatic solid tumors

DETAILED DESCRIPTION:
The goal of this clinical trial is to test patients with locally advanced or metastatic solid tumors. The main questions it aims to answer are:

* To evaluate the safety and tolerability of SM3321 in patients with locally advanced or metastatic solid tumors.
* To determine dose-limiting toxicities (DLTs) , Maximum tolerated dose(MTD) and Recommended phase 2 dose (RP2D)of SM3321 in the treatment of patients with locally advanced or metastatic solid tumors. .
* To evaluate the Pharmacokinetics (PK) profile of SM3321 in patients with locally advanced or metastatic solid tumors after single and multiple administration.
* To evaluate the immunogenicity of single and multiple administration of SM3321 in patients with locally advanced or metastatic solid tumors.
* To evaluate the initial antitumor activity of SM3321 in patients with locally advanced or metastatic solid tumors.
* To further evaluate serum biomarkers and explore the potential relationship between these markers and the antitumor activity and safety of SM3321.
* To explore the relationship between dose and/or PK exposure and effects(including anti-tumor activity and safety).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older.
2. Subjects with histologically or cytologically confirmed unrespectable locally advanced or metastatic solid tumors.
3. The subject's disease progresses after receiving adequate standard treatment or is intolerant to standard treatment or has no effective standard treatment options available.
4. Subjects in this study must have at least one evaluable lesion (based on RECIST v1.1).
5. Expected survival ≥12 weeks
6. ECOG PS score 0-2 points
7. The function of the major organs is basically normal, and the laboratory examination within 7 days or less before the first administration meets the following standards:

   a) Liver function:
   * AST/ALT ≤ 2.5 × ULN (ULN= upper limit of normal);If liver metastasis occurs, AST/ALT≤5×ULN;
   * Serum total bilirubin ≤ 1.5 × ULN;Or in cases of Gilbert syndrome ≤3×ULN; b) Blood routine (no hematopoietic growth factor or blood transfusion was used within 2 weeks before enrollment) :
   * Hemoglobin ≥ 90 g/L;
   * Platelet count ≥100×10^9/L;
   * Absolute neutrophil count ≥1.5×10^9/L. c) Kidney function:
   * Creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula). d) Coagulation function:
   * International normalized ratio (INR) ≤1.5×ULN.
8. Female subjects of reproductive age must have a negative blood pregnancy test within 3 days prior to the first use of the study drug; Eligible subjects (men and women) who are fertile (defined as sexually mature and biologically fertile) must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence, etc.) with their partner during the study period and for at least 6 months after the last dose.
9. Willing to participate in clinical research, understand and sign informed consent, and follow up and abide by research procedures on time.

Exclusion Criteria:

1. Known allergy to SM3321 or its formulation components.
2. Previously received the following anti-tumor therapy:

   1. Chemotherapy, targeted therapy, immunotherapy, or other anticancer therapy within 28 days or 5 half-lives (whichever is shorter) prior to initial administration of the investigational therapy, except for the following:

      * anti-programmed death receptor-1 / programmed death receptor-ligand 1 antibodies used within 1.5 months;
      * nitrosourea or mitomycin eluting period ≤6 weeks;
      * Washout period of fluoropyrimidine or small molecule targeted drugs ≤5 half-lives or 2 weeks (whichever is longer);
      * The washout period for herbal treatments with anticancer indications is ≤2 weeks.
   2. Radiotherapy received within 4 weeks prior to the first dosing of the study treatment, allowing a single fractionated radiotherapy for symptom relief.
   3. The subject has participated in any other clinical study and received the trial drug within 28 days prior to the first administration of the study drug.
3. Major surgery within 28 days before dosing or major surgery expected during the study period.
4. There was acute toxicity from prior antitumor therapy that had not returned to ≤ grade 1 or baseline levels specified by the inclusion criteria prior to first administration (based on NCI-CTCAE v5.0).
5. Uncontrolled or severe cardiovascular disease, including but not limited to any of the following:

   1. Prolonged QTc (using Fridericia's correction formula), male >450 ms/ female >470 ms, or congenital long QT syndrome;
   2. Left ventricular ejection fraction (LVEF) <50% was assessed by Multiple-gated acquisition (MUGA) or ECHO;
   3. any of the following in the 6 months prior to screening: > Grade 2 ventricular arrhythmia, severe/unstable angina, congestive heart failure (New York heart association (NYHA) III orGrade IV), coronary artery bypass grafting, myocardial infarction, cerebrovascular accident, or transient ischemic attack;
   4. Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg).If blood pressure can be controlled within the above limits by antihypertensive therapy, subjects with a history of hypertension will be admitted to the study.,
6. Concurrent history of severe chronic or active infection:

   1. The subject has active hepatitis B, defined as:If HepatitisB surface antigen (HBsAg) is positive, hepatitisB virus (HBV) Deoxyribonucleic acid (DNA) should be tested for HepatitisB virus (HBV).HBV DNA was higher than the lower limit of quantitative value.
   2. The subject has active Hepatitis C, defined as: if Hepatitis C virus (HCV) antibodies are positive, HCV Ribonucleic acid (RNA) should be tested, and HCVRNA is positive;
   3. Known to have Acquired immune deficiency syndrome (AIDS) or Human immunodeficiency viru (Human immunodeficiency viru)Hiv-infected subjects may be eligible for study participation if the CD4+ T cell count is ≥350 cells /µL and there is no history of opportunistic infection as defined by AIDS.
   4. other severe chronic infections, including but not limited to hospitalization for infectious complications, bacteremia, severe pneumonia, or active tuberculosis complications, within 4 weeks prior to initial administration of SM3321;Or an uncontrolled active infection or unexplained fever >38 ° C occurred within 7 days prior to first administration of SM3321.
7. Uncontrolled co-morbidities such as:

   1. Subjects with known active primary tumors or metastases of the Central nervous system (CNS);Note: Subjects with previously treated primary CNS tumors/metastases may participate in the study, provided that they are clinically stable for at least 2 weeks, have no evidence of new BMS or BMS enlargement, and were first dosed with SM3321 The steroid dose was not increased during the first 14 days to manage CNS symptoms.Subjects with cancerous meningitis or pia spread or spinal cord compression were excluded from this study even if clinically stable.
   2. known to have other malignancies that are currently advanced or have required aggressive treatment within the past 5 years (except for non-melanoma skin basal cell carcinoma or squamous cell carcinoma, breast/cervical carcinoma in situ, superficial bladder carcinoma and other in situ cancers that have been treated radically and have no evidence of disease recurrence);
   3. A history of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to enrollment;
   4. Significant malnutrition, such as the need for intravenous nutritional solutions. Patients with stable malnutrition for more than 4 weeks after correction before the first dose of the study drug could be enrolled;
   5. Other acute or chronic medical conditions or abnormalities in laboratory testing that may increase the risks associated with participation in the study or use of the study product, or interfere with the interpretation of the study results and, in the judgment of the investigator, render the subject ineligible for participation in the study.
8. Pregnant or lactating women.
9. Have a history of active autoimmune disease, such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, or have received long-term systemic steroid therapy (at doses greater than 10 mg prednisone daily equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first administration of the study drug. Exceptions include: clinically stable autoimmune thyroid disease; Receive inhaled or topical corticosteroid therapy, such as intraocular, intraarticular, and intranasal administration of prednisone equivalent ≤10 mg daily; Short-term use of corticosteroids (no more than 7 days) for preventive treatment (for example, to prevent hypersensitivity to contrast agents or non-autoimmune allergic diseases);As well as replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes, physiocorticoid replacement for adrenal or pituitary insufficiency).
10. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
11. Received systemic immunomodulatory drugs, such as thymosin, IL-2, and IFN, within 14 days prior to the first administration of the study drug.
12. People who have a clear history of mental disorders and take medication for treatment.
13. People with a history of drug abuse or use.
14. Receive or will receive live vaccine within 30 days prior to the first dose of the study drug, or plan to receive any live vaccine during the study.
15. The Investigator believes that the subject may have other factors that could affect the study results and interfere with the subject's participation in the overall study process, including previous or existing medical conditions, abnormal treatments or laboratory tests, and the subject's unwillingness to comply with all procedures, study restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | DLT observation period: 28 days after the first dose [i.e., 1 Cycle ]
  The highest dose when the proportion of subjects with DLT events during the DLT observation period was less than 1/3 or 2/6 of
Phase II recommended dose（RP2D) | DLT observation period: 28 days after the first dose [i.e., 1 Cycle ]
  RP2D will be determined based on safety, tolerability, PK, and PD study results, and may be at MTD/MAD or lower dose levels.
  The RP2D cohort will include at least six evaluable subjects to further clarify safety and tolerability.
  Adverse events in subjects that meet the definition of DLT outside the DLT observation period will not be used as a basis for dose escalation, but will be used as a reference for subsequent dose design and for evaluating the overall safety of future recommended doses
Safety evaluation-1 | Screen Period(Day-28~Day-1),Cycle 1 (Day1, 2, 3, 4, 6, 8, 15,22, 23, 24, 25,27） (Cycle 2~Cycle N) Day 1±3 Days, within 7 days after stop dosing, 30±5 days after last dosing, 90±5 days after last dosing (1 Cycle=28 Days)
  Incidence and severity of DLT, adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE)(evaluated per [National Cancer Institute-Common Terminology Criteria for Adverse Events，NCI-CTCAE] v5.0)
Safety evaluation-2 | Screen Period(Day-28~Day-1),Cycle 1 (Day1, 8, 15,22） (Cycle 2~Cycle N) Day 1±3 Days, within 7 days after stop dosing, 30±5 days after last dosing, 90±5 days after last dosing (1 Cycle=28 Days)
  Clinically significant abnormalities in laboratory tests, including blood routine examination, coagulation function, blood biochemistry, urine analysis, viral serology
Safety evaluation-3 | On the day of dosing, within 1 hour before dosing, every 15±5 minutes during dosing, at the end of dosing (within 5 minutes), and every 30±5 minutes after dosing. within 4 hours after the end of the first dosing
  vital signs, including respiratory rate, heart rate, body temperature and blood pressure
Safety evaluation-4 | Screen Period(Day-28~Day-1),Cycle 1 (Day1, 8, 15,22） (Cycle 2~Cycle N) Day 1±3 Days, within 7 days after stop dosing, 30±5 days after last dosing, 90±5 days after last dosing (1 Cycle=28 Days)
  physical examination, examination of the entire human system/organ (skin, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, respiratory, cardiovascular, gastrointestinal, limbs, abdomen, back, musculoskeletal, nervous system and mental state)
Safety evaluation-5 | Within 1 hour before dosing, 30 minutes after ending dosing, and 30 minutes after starting dosing 4 hours
  electrocardiogram (ECG)
Safety evaluation-6 | Scans or examinations are performed during the screening period and when clinically indicated
  echocardiography (ECHO)
Safety evaluation-7 | Screen Period(Day-28~Day-1), (Cycle 2~Cycle N) Day 1±3 Days, within 7 days after stop dosing (1 Cycle=28 Days)
  physical status (PS) in the Eastern United States Oncology Consortium (ECOG)

CONTACTS AND LOCATIONS:
Overall Officials: Qi Li, Dr., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The second affiliated hospital Zhejiang university School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No